CLINICAL TRIAL: NCT01705717
Title: Treatment Outcomes in the Management of Patients With Chronic Hepatitis C: A Case Study of Faculty of Medicine Vajira Hospital, University of Bangkok Metropolis
Brief Title: A Retrospective Study of Real World Treatment Outcomes of Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25436
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- cohort

SUMMARY:
This retrospective, observational study will assess the real world treatment out comes in the management of patients with chronic hepatitis C. No prospective ass essment or procedure with patients during this study will be conducted. Data wil l be collected from patient medical records of the year 2000-2011.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with chronic hepatitis C during the year 2000 to 2010
* Availability of data for at least 6 months following the diagnosis date

Exclusion Criteria:

* Patients who participated in an investigational clinical trial
* Co-infection with hepatitis A, hepatitis B, hepatitis D, and/or human immunodeficiency virus (HIV)
* Patients with known severe medical conditions that are contraindicated to HCV treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective survey of medical records of patients with chronic hepatitis C
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Faculty of Medicine Vajira Hospital; Division of Gastroenterology and Hepatology, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Cirrhotic Chronic Hepatitis C (CHC) Observation Only: Participants with newly diagnosed during the years 2000 through 2010 non-cirrhotic CHC and related morbidities were treated per the standard of care or local clinical practice and at the discretion of the physician for up to 36 months.
- Hepatitis C Virus (HCV) - Related Cirrhosis Observation Only: Participants with newly diagnosed during the years 2000 through 2010 HCV-related compensated cirrhosis and related morbidities were treated per the standard of care or local clinical practice and at the discretion of the physician for up to 36 months.
Period: Overall Study
Arm/Group | Non-Cirrhotic Chronic Hepatitis C (CHC) Observation Only | Hepatitis C Virus (HCV) - Related Cirrhosis Observation Only
Started | 37 | 12
Completed | 35 | 7
Not Completed | 2 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Non-Cirrhotic CHC Observation Only: Participants with newly diagnosed during the years 2000 through 2010 non-cirrhotic CHC and related morbidities were treated per the standard of care or local clinical practice and at the discretion of the physician for up to 36 months.
- HCV - Related Cirrhosis Observation Only: Participants with newly diagnosed during the years 2000 through 2010 HCV-related compensated cirrhosis and related morbidities were treated per the standard of care or local clinical practice and at the discretion of the physician for up to 36 months.
- Total: Total of all reporting groups
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only | Total
Number analyzed (Participants) | 37 | 12 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (10.9) | 53.9 (8.2) | 47.2 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 25 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR): Percentage of Participants Who Were HCV Seronegative at 6 Months After Completing Therapy
Description: SVR was defined a negative result upon polymerase chain reaction (PCR) ribonucleic acid (RNA) diagnostic testing after 6 months of treatment.
Time Frame: 6 months
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only
Number analyzed (Participants) | 37 | 12
percentage of participants | 59.5 | 58.3

2. Secondary Outcome: Percentage of Participants Who Were HCV Seronegative at the End of Treatment
Description: End-of-treatment response (ETR) was defined as a negative result upon PCR RNA diagnostic testing at the end of treatment.
Time Frame: End of Study, up to 36 months after diagnosis.
Population: All enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only
Number analyzed (Participants) | 37 | 12
percentage of participants | 91.9 | 91.6

3. Secondary Outcome: Percentage of Participants With HCV Relapse (Biochemical or Virological) After Treatment Completion
Description: HCV relapse was determined by PCR RNA diagnostic testing. Virological relapse was defined as subsequent reappearance of serum HCV RNA after completion of therapy in participants who achieved end of treatment virological response (undetectable HCV RNA). Biochemical relapse was defined as subsequent rise in serum alanine aminotransferase (ALT) level after end of treatment with normal ALT.
Time Frame: End of Study, up to 36 months after diagnosis.
Population: All enrolled participants;
Measure: Number; unit: percentage of participants
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only
Number analyzed (Participants) | 22 | 7
percentage of participants
  Virological Relapse | 0 | 0
  Biochemical Relapse | 0 | 14.3

4. Secondary Outcome: Percentage of Participants Who Progressed From CHC to Cirrhosis
Time Frame: Diagnosis and End of Study, up to 36 months after diagnosis.
Population: All enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only
Number analyzed (Participants) | 37 | 12
percentage of participants | 0 | 0
Statistical Analysis 1: Comparison: Non-Cirrhotic CHC Observation Only vs HCV - Related Cirrhosis Observation Only; Test type: Superiority or Other; p = 0.034, Chi-squared

5. Secondary Outcome: Percentage of Participants Who Progressed From CHC to Hepatocellular Carcinoma (HCC)
Time Frame: Diagnosis and End of Study, up to 36 months after diagnosis.
Population: All enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only
Number analyzed (Participants) | 37 | 12
percentage of participants | 2.7 | 8.3
Statistical Analysis 1: Comparison: Non-Cirrhotic CHC Observation Only vs HCV - Related Cirrhosis Observation Only; Test type: Superiority or Other; p = 0.007, Chi-squared

6. Secondary Outcome: Percentage of Participants Who Died
Description: Any cause of death (including non-liver disease related) was reported.
Time Frame: Diagnosis and End of Study, up to 36 months after diagnosis
Population: All enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Non-Cirrhotic CHC Observation Only | HCV - Related Cirrhosis Observation Only
Number analyzed (Participants) | 37 | 12
percentage of participants | 2.7 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the begininng of treatment through the end of the study, approximately 36 months. This was a retrospective analysis study; safety reporting was generated spontaneously by physician discretion.
Description: All participants for whom safety data was collected are included in the safety analysis. Systematic collection of safety data was not mandatory according to the protocol.
Groups:
- All Participants: Participants with newly diagnosed during the years 2000 through 2010 non-cirrhotic CHC or HCV-related compensated cirrhosis and related morbidities were treated per the standard of care or local clinical practice and at the discretion of the physician for up to 36 months.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 4/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=47)
Anemia (Blood and lymphatic system disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Intracranial hemorrhage (Vascular disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Severe anemia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.